CLINICAL TRIAL: NCT04229563
Title: PATHFINDER I: Post-Market Registry of AURYON™ Atherectomy Device in Subjects Affected With Infrainguinal Peripheral Artery Disease (PATHFINDER-Registry, EX-PAD-05)
Brief Title: Post-Market Registry of AURYON™ Atherectomy Device in Subjects Affected With Infrainguinal Peripheral Artery Disease
Acronym: PATHFINDER-I
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EX-PAD-05
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Infrainguinal Peripheral Artery Disease; Peripheral Arterial Disease; PAD
Keywords: Peripheral Artery Disease; Peripheral Occlusive Disease; Peripheral Artery Stenonsis; Artery Restenosis; Arterial Occlusive Disease; Peripheral Vascular disease; Laser recanalization; Endovascular treatment or Procedure or Surgery; Calcified Lesions; Atherectomy; Intermittent Claudication; Claudication pain; Arterial Calcification; Critical Limb Ischemia; CLI; Acute Limb Ischemia; Acute Arterial Occlusion; Infra-inguinal Stenosis or Occlusion; Femoral Artery Stenosis; Femoral-Popliteal Arterial Disease; Tibial Stenosis; In-stent Restenosis; Stenotic lesion; Peripheral Artery Revascularization; Lower Limb Arterial Calcification; Laser-assisted angioplasty; Above the Knee calcification; ATK Calcification; Below the Knee Calcification; Chronic total occlusion; CTO; Superficial Femoral Artery Disease; Target Lesion revascularization; Atherectomy Catheter; Observational Study; Registry; Walking Impairment questionnaire; Intravascular ultrasound; Ankle-Brachial Pressure Index; Toe-Brachial Index; Rutherford Classification; ABI; TBI; Peak Systolic Velocity Ratio; Auryon System; Eximo Medical; AngioDynamics; B-Laser; Real World Evidence
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases; Peripheral Vascular Diseases; Intermittent Claudication; Chronic Limb-Threatening Ischemia; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study patients: Eligible PAD patients who are routinely treated with atherectomy by AURYON™ Atherectomy System.
  Interventions: Device: AURYON™ System

INTERVENTIONS:
Device: AURYON™ System — The AURYON™ System consists of two sub-units: 1) a single use catheter ("AURYON™ catheter"); and 2) a laser system.

SUMMARY:
The PATHFINDER I Registry is a prospective, non-randomized, single arm, multicenter observational study. It is a pilot registry study towards a subsequent large pivotal phase registry. This pilot registry is aimed to evaluate the performance (peri-procedural) and clinical outcomes (intermediate and long-term) of the AURYON™ Atherectomy System, within the initial launch phase of the product in the market.

DETAILED DESCRIPTION:
US multicenter, prospective, single-arm, observational post market Registry. A pilot registry towards a subsequent large pivotal registry (PATHFINDER II), aimed to evaluate the safety and efficacy of Auryon™ Atherectomy System in the treatment of de novo, re-stenotic and ISR lesions in infra-inguinal arteries of Peripheral Artery Diseases (PAD) subjects, in a real-world setting within the initial launch phase of the product in the market.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. Subject is a candidate for atherectomy for infra-inguinal peripheral artery disease.
3. Documented symptomatic atherosclerotic peripheral artery disease with claudication or critical limb ischemia (CLI) (Rutherford Classification 2-5 ).
4. Subject is capable and willing to comply with the scheduled follow up
5. Subject is able and willing to sign a written Informed Consent Form (ICF).

Exclusion Criteria:

1. Target lesion is in an arterial bypass.
2. Planned use of another atherectomy device in the same procedure
3. Co-morbid condition(s) with less than 1yr anticipated survival that could limit the subject's ability to participate in the trial or to comply with follow-up requirements or impact the scientific integrity of the study.
4. Participating in another study on an interventional non-cleared device, that could impact the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infra-inguinal PAD undergoing atherectomy with the AURYON™ Atherectomy System.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2023-04-17 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy: Acute Procedural Success | Peri-procedural (by the end of the index procedure)
  Percentage of subjects with successful revascularization of target vessel defined as ≤30% residual stenosis at the index lesion post AURYON™ atherectomy and final adjunctive treatment (if required), as evaluated by angiographic corelab.
Primary Safety: Freedom from Peri-procedural major adverse events (PPMAE) | Till discharge, an average of 5 days
  Percentage of subjects with freedom from peri-procedural major adverse events (PPMAE), defined as (a) flow-limiting dissection, (b) clinically significant distal embolization, (c) bailout stenting, (d) major/unplanned amputation, (e) target vessel perforation requiring endovascular or surgical repair or (f) death, till discharge.

SECONDARY OUTCOMES:
Rate of device related complications requiring intervention | Till discharge, an average of 5 days
  Rate of device related complications requiring intervention, defined as peri procedural MAEs, reported by the operating physician as caused directly due to the use of the AURYON device.
Rates of MAEs over time | Post-discharge (at 30-days, 6-, 12-, and 24-months)
  Rates of post-discharge MAEs over time; defined as: (a) Unplanned target limb amputation, (b) cardiovascular death, (c) clinically driven target lesion revascularization , (d) target vessel revascularization (TVR).
Patency rate | Post-discharge (at 6-, 12-, and 24-months)
  Patency rate, defined as <50% stenosis at the treated lesion, with peak systolic velocity ratio (PSVR) of <2.5, as assessed quantitatively by Duplex ultrasonography (DUS) performed in a lab that achieved Vascular Laboratory Accreditation, at 6, 12, and 24 months.
Occlusion freedom | Post-discharge (at 6-, 12-, and 24-months)
  Only for BTK lesions: freedom from occlusion (100% stenosis by DUS) combined with freedom from CD-TLR
Clinical outcome 1 - ankle brachial index (ABI) | Post-discharge (at 6-, 12-, and 24-months)
  Change in ankle brachial index (ABI or TBI if needed) at 6, 12, and 24, months, compared to baseline.
  Ankle-Brachial Index (ABI) si an ankle/arm blood pressure ratio. Normal value ranges between 0.9-1.3. Under 0.9 index means blood has a difficult time getting to legs & feet; 0.4-0.9 indicates mild-moderate PAD; 0.4 and lower indicates severe PAD. Positive difference between time-points represents a clinical improvement through time and vice versa.
Clinical outcome 2 - walking impairment questionnaire (WIQ) | Post-discharge (at 6-, 12-, and 24-months)
  Change in walking impairment questionnaire (WIQ) score at 6, 12, and 24, months, compared to baseline.
  WIQ is a patient fulfilled survey to grade physical ability representing PAD progress, has 3 sub-scales (walking speed, distance, climbing stairs), when the total score ranges between 0-100, higher value = better outcome. Positive difference between time-points represents a clinical improvement through time and vice versa.
Clinical outcome 3 - Rutherford clinical categories (RCC) | Post-discharge (at 6-, 12-, and 24-months)
  Change in Rutherford clinical category at 6, 12, and 24, months, compared to baseline.
  Rutherford Classification is a doctor determined 7 stages scale (0= Asymptomatic, 6= Severe ischemic ulcers/frank gangrene) representing PAD progress, lower value = better outcome. Positive difference between time-points represents a clinical deterioration through time and vice versa.

OTHER OUTCOMES:
Exploratory endpoint: IVUS | Peri-procedural (by the end of the index procedure)
  Intravascular ultrasound assessment pre- and post-Auryon and correlation with angiographic findings (e.g. lesion length, MLA -minimal lumen area gain, calcium severity and removal, etc.). This endpoint will be analyzed only for cases that used IVUS as a routine practice in the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: TBD TBD, Study Chair
Locations (5):
- United States (5):
  - Pulse Cardiovacular, Scottsdale, Arizona
  - Pima Vascular, Tucson, Arizona
  - Comprehensive Cardiovascular, Davenport, Florida
  - Midwest Cardio. research foundation, Davenport, Iowa
  - Hurricane Cardiology, New Braunfels, Texas

REFERENCES:
- [Derived] Das TS, Shammas NW, Yoho JA, Martinez-Clark P, Ramaiah V, Leon LR, Pacanowski JP, Tai Z, Ali V, Arslan B, Rundback J. Solid state, pulsed-wave 355 nm UV laser atherectomy debulking in the treatment of infrainguinal peripheral arterial disease: The Pathfinder Registry. Catheter Cardiovasc Interv. 2024 May;103(6):949-962. doi: 10.1002/ccd.31023. Epub 2024 Apr 2. PMID 38566525